CLINICAL TRIAL: NCT06815653
Title: Digital Intervention for Psychedelic Preparation (DIPP): A Randomised Controlled Feasibility Trial Comparing Meditation and Music-Based Programs in Healthy Volunteers.
Brief Title: Digital Intervention for Psychedelic Preparation (DIPP): Comparing Meditation and Music-Based Programs
Acronym: (DIPP-RCFT)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19113/003
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: psilocybin; meditation; preparation; digital
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a meditation-based preparation group or a music-listening control group. Both groups will engage in their assigned activity daily for 21 days leading up to a single psilocybin session, where they will each receive a 25 mg oral dose of psilocybin.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meditation (Experimental): Digital Intervention for Psychedelic Preparedness (DIPP) (Meditation) - A 21-day self-guided digital intervention based on four validated preparedness factors (Knowledge-Expectation, Psychophysical-Readiness, Intention-Preparation, and Support-Planning) (McAlpine et al., 2024). Participants will access a digital platform daily, completing structured, guided meditation sessions that progressively introduce and develop meditation techniques. The program includes daily mood assessments, journaling exercises, and weekly module-specific tasks.
  Interventions: Drug: Psilocybin 25mg
- Music Listening (Active Comparator): Digital Intervention for Psychedelic Preparedness (DIPP) (Music-listening control) - Identical to the meditation arm in duration, structure, and theoretical framework, but participants engage in music-listening sessions using the same background music as the meditation arm, without guided meditation instructions. All other components (mood assessments, journaling, weekly tasks) remain the same.
  Interventions: Drug: Psilocybin 25mg

INTERVENTIONS:
Drug: Psilocybin 25mg — Psilocybin PEX010 is an investigational drug provided in capsule form, containing a 25 mg dose of synthetic psilocybin. The product is manufactured under Good Manufacturing Practice (GMP) standards to ensure purity, potency, and consistency. Each participant will receive a single oral dose of 25 mg psilocybin in a hydroxypropyl methylcellulose (HPMC) capsule. The intervention is administered once during the study session, with the effects expected to last approximately 4 to 6 hours.

SUMMARY:
This randomised controlled feasibility trial evaluates the Digital Intervention for Psychedelic Preparation (DIPP), a novel 21-day self-guided program designed to prepare individuals for psychedelic experiences. Forty healthy volunteers will be randomly assigned to either a meditation-based intervention or a music-based control condition. Both groups will follow identical program structures, with the key distinction being their daily practice focus: meditation or music listening. Following the 21-day preparation period, participants will undergo a supervised 25 mg psilocybin session at University College London. Assessment visits include an in-person follow-up at 2 weeks post-session, followed by online assessments at 3, 6, and 9 months. The primary outcomes include operational feasibility (recruitment rates and participant retention) and intervention adherence (completion rates of DIPP program activities). Secondary outcomes include participant ratings of the platform's feasibility, acceptability, and usability, as well as changes in psychedelic preparedness, the quality of the psychedelic experience, and mental wellbeing over time.

DETAILED DESCRIPTION:
Growing evidence demonstrates the therapeutic potential of psychedelic substances, particularly psilocybin, in addressing mental health challenges and enhancing psychological well-being. While psychedelic experiences can catalyse profound positive changes, they can also be psychologically challenging and potentially destabilising, underscoring the need for thorough preparation. Studies consistently show that an individual's psychological state prior to psychedelic administration significantly influences both the acute experience and its lasting benefits. However, structured preparation protocols designed to optimise this pre-psychedelic state remain understudied despite their crucial role in therapeutic outcomes.

Digital health interventions offer a promising solution for delivering standardised preparation protocols at scale. Meditation-based approaches warrant particular investigation, as they systematically cultivate both immediate psychological states and enduring traits (e.g. non-judgemental acceptance) beneficial for psychedelic experiences. Through regular practice, meditation promotes trait-like metacognitive awareness, emotional regulation, and tolerance of uncertainty - qualities particularly valuable for navigating altered states of consciousness. These benefits are supported by neuroscientific evidence showing that meditation and psychedelics influence similar brain networks and mechanisms. While traditional meditation training often requires substantial time investment and in-person instruction, digital platforms can provide efficient structured guidance without the need for face-to-face support from a trained instructor, while maintaining essential elements of practice. This combination of accessibility and evidence-based benefits makes digital meditation platforms particularly well-suited for preparing individuals for psychedelic experiences.

This randomised controlled feasibility trial evaluates the Digital Intervention for Psychedelic Preparation (DIPP), a 21-day self-guided program. Forty healthy volunteers will be randomised 1:1 to either a meditation-based intervention or music-based control condition. Both groups will engage with identical program structures, differing only in their daily practice (meditation versus music listening). Following preparation, all participants will undergo a supervised 25 mg psilocybin session at University College London, with follow-up assessments conducted in person at 2 weeks and online at 3, 6, and 9 months post-intervention.

The primary outcomes address two key aspects of feasibility: operational feasibility and intervention adherence. Operational feasibility evaluates study-wide metrics, including recruitment efficiency (target ≥1 participant per week) and participant retention (target ≥70% completion through the 2-week post-dose follow-up). Intervention adherence focuses on participant engagement with the DIPP activities (meditation or music listening), assessed through completion rates for daily sessions, mood check-ins, journal entries, and weekly tasks, with a target of ≥70% of participants achieving an average completion rate of 70% or higher. Secondary outcomes, reported descriptively for both conditions, include implementation measures such as subjective feasibility (SFIS), acceptability (TFA), and usability (SUS/MARS) ratings. Efficacy measures assess changes in psychedelic preparedness (PPS) from baseline to post-DIPP intervention, the qualities of the acute psychedelic experience (11-Dimensional Altered States of Consciousness Scale [11D-ASC] and Challenging Experience Questionnaire [CEQ]) following dosing, and changes in mental wellbeing (Warwick-Edinburgh Mental Wellbeing Scale [WEMWBS]) from baseline through the 2-week post-dose follow-up.

As such, this study will investigate the feasibility of implementing a digital preparation protocol within a research setting, while gathering preliminary data on engagement, acceptability, and potential efficacy. The findings will inform refinements to the DIPP platform and protocol, supporting the development of accessible, standardised preparation methods for psychedelic research and therapy as the field continues to expand into diverse clinical and community-based settings.

ELIGIBILITY:
Inclusion Criteria:

Aged 21-65 years. Limited psychedelic use (0-5 sessions involving a high/full dose, defined as producing noticeable psychoactive effects beyond microdosing; none in the past 6 months).

Minimal meditation experience (≤10 sessions exceeding 30 minutes; no retreats or regular practice).

Native English speaking. Normal or corrected-to-normal colour vision. Able and willing to provide informed consent. Able to engage with all study requirements, including in-person and remote sessions.

UK resident registered with a primary care practice. Agree to allow research team contact with primary/secondary care teams if needed.

Access to mobile smartphone.

Exclusion Criteria:

Current or past psychiatric diagnosis (e.g., depression, anxiety) unless in clear remission for at least 5 years and assessed as low-risk.

Current or past psychotic or bipolar disorder diagnosis. First degree relative with psychotic or bipolar disorder diagnosis. Current or past behaviours, including attempts, planning or intention. Medically significant physical health conditions (e.g., cardiovascular disease, uncontrolled hypertension, epilepsy, migraines, focal scalp sensitivity, or any condition posing a safety risk).

Use of medications interacting with psilocybin (e.g., antipsychotics, SSRIs, SNRIs, TCAs, mood stabilisers).

Psychoactive drug use within 30 days (except nicotine or caffeine). Pregnancy, planning pregnancy, or breastfeeding. Participation in a drug trial within 6 months. MRI contraindications (e.g., metal implants, pacemakers, severe claustrophobia).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment efficiency | Assessed at Visit 4 (2 weeks post-dose)
  Weekly rate of participant enrollment and randomisation. Success is defined as ≥1 participant per week (average) until target sample (N=40) achieved
Study retention | Assessed at Visit 4 (2 weeks post-dose)
  Percentage of randomised participants completing the 2-week post-dose follow-up assessment. Success is defined as ≥70% completion rate
DIPP intervention adherence | Assessed at Visit 2 (1 day pre-dose)
  Task completion rates across three daily tasks (meditation/music practice, mood rating, journal entry) and two weekly tasks. Success is defined as ≥70% of participants achieving an average completion rate of ≥70% across all required tasks

SECONDARY OUTCOMES:
DIPP platform feasibility as measured by the Subjective Feasibility of Intervention Scale (SFIS) | Administered at Visit 2 (1 day pre-dose)
  The Subjective Feasibility of Intervention Scale (SFIS) measures perceived practicality, resource demands and integration into existing workflows of the DIPP protocol. Possible scores range from 9 to 45, with higher scores indicating better feasibility
DIPP platform acceptability as measured by the Theoretical Framework of Acceptability Scale (TFA) | Administered at Visit 2 (1 day pre-dose)
  The Theoretical Framework of Acceptability Scale (TFA) measures perceived appropriateness and satisfaction with the DIPP platform. Possible scores range from 7 to 35, with higher scores indicating better acceptability
DIPP platform usability and engagement as measured by the System Usability Scale (SUS) and Mobile Application Rating Scale (MARS) | Administered at Visit 2 (1 day pre-dose)
  The System Usability Scale (SUS) and Mobile Application Rating Scale (MARS; functionality and aesthetics subscales only) measure platform user-friendliness and app quality respectively. Combined scores range from 16 to 80, with higher scores indicating better usability/engagement
Psychedelic Preparedness as measured using the Psychedelic Preparedness Scale (PPS) | Administered at Visit 1 and 2 (1 day pre-dose)
  Between-group differences in psychedelic preparedness will be assessed using the Psychedelic Preparedness Scale (PPS), a validated 20-item self-report measure. The PPS evaluates four domains: knowledge-expectation, psychophysical-readiness, intention-preparation, and support-planning. Individual total scores (range: 20-140) and mean factor scores (range: 1-7) will be calculated, with higher scores indicating greater preparedness
Positive quality of acute psychedelic experience as measured by the Altered States Consciousness Questionnaire (11D-ASC) | Administered at Visit 3 (8 hours post-dose)
  The Altered States Consciousness Questionnaire (11D-ASC) measures the subjective effects of the psychedelic experience. To assess the positive quality of the experience, this study will focus on the Oceanic Boundlessness (OBN) factor to assess participants' subjective experience of unity, boundary dissolution, and interconnectedness during the psilocybin session. Possible standardised scores range from 0 to 1, with higher scores indicating a more positive quality of acute psychedelic experience.
Challenging psychological experience during the psychedelic experience as measured by the Challenging Experience Questionnaire (CEQ) | Administered at Visit 3 (8 hours post-dose)
  The Challenging Experience Questionnaire (CEQ) measures various aspects of challenge experienced during a psychedelic experience. To assess challenging psychological experiences during the psilocybin session, this study will focus on the combined mean score on four CEQ subscales (Fear, Insanity, Isolation, and Paranoia). Possible scores range from 0 to 5, with higher scores indicating a more challenging psychedelic experience
Mental wellbeing as measured by the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Administered at Visit 1, 2, 3 and 4 (2 weeks post-dose)
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) measures psychological functioning and emotional wellbeing. Possible scores range from 14 to 70, with higher scores indicating better wellbeing

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying published results will be shared. This includes questionnaire responses, behavioural task data, hormonal measures, EEG and ECG recordings. Access to these data will be granted upon reasonable request to the corresponding author, subject to a data-sharing agreement ensuring participant confidentiality and compliance with data protection regulations. De-identified fMRI data will be made publicly available in suitable repositories, where permitted by institutional policies and applicable regulations. Requests will be evaluated based on the scientific merit of proposed analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be available beginning 6 months after publication of the primary results and will remain available for 5 years. De-identified fMRI data will be deposited in a public repository as soon as institutional approvals permit. Other de-identified data (questionnaire, behavioural, hormonal, EEG, and ECG) and analytic code will be shared upon reasonable request to the corresponding author within this period, subject to a data-sharing agreement.
Access Criteria: Qualified researchers affiliated with academic or healthcare institutions may request access to de-identified IPD and supporting information for scientifically sound, ethically approved analyses that align with the study's objectives. Requests must include a detailed research proposal, analysis plan, and evidence of ethical approval or exemption. Proposals will be reviewed by the study's data access committee to assess scientific merit, feasibility, and compliance with participant confidentiality. Approved users must sign a data-sharing agreement. Requests should be submitted via email to the corresponding author.